CLINICAL TRIAL: NCT06122987
Title: An Open-label, Single-arm, Single-center Study Evaluating the Hemodynamic Response to Angiotensin-II When Used as the Second Vasopressor Agent for Septic Shock
Brief Title: Hemodynamic Response to Angiotensin-II When Used as the Second Vasopressor Agent for Septic Shock
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kingman Regional Medical Center (Other)
Collaborators: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Principal Investigator, Tyson Dietrich, Pharmacist, Kingman Regional Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRMC 0284
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Septic Shock; Shock; Sepsis; Systemic Inflammatory Response Syndrome
Keywords: Sepsis; Angiotensin II; Hydrocortisone
MeSH Terms: conditions — Shock, Septic; Shock; Sepsis; Systemic Inflammatory Response Syndrome | interventions — Angiotensin II; Hydrocortisone; Giapreza

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single Arm (Experimental): Drug: Angiotensin II Other Names: Giapreza
  Interventions: Drug: Angiotensin II and hydrocortisone sodium succinate

INTERVENTIONS:
Drug: Angiotensin II and hydrocortisone sodium succinate — Intravenous infusion angiotensin II (titrated for each individual patient by effect) and hydrocortisone 50 mg intravenous bolus every 6 hours.
  Other Names: Giapreza

SUMMARY:
Norepinephrine is a catecholamine that is the first-line vasopressor for septic shock. The addition of non-catecholamine vasopressors, including vasopressin and angiotensin-II may be used in adults with septic shock that have inadequate mean arterial pressure while on norepinephrine. Uncertainty exists regarding the timing of initiation of these agents and there is a lack of data comparing their safety and efficacy.

The current literature suggests that earlier initiation of angiotensin-II will have a more significant reduction on norepinephrine-equivalent dose compared to later initiation. In addition, approximately half of patients initiated on vasopressin do not have an early hemodynamic response 6 hours after initiation. The purpose of this study is to evaluate the efficacy of angiotensin-II when used as the second vasopressor agent for septic shock.

DETAILED DESCRIPTION:
Objectives:

Primary Objective:

1. To evaluate the efficacy of ang-II when used as the second vasopressor agent for septic shock

Secondary Objectives:

1. To assess the duration of response to ang-II
2. To assess overall survival
3. To assess the amount of time spent in the ICU
4. To assess the need for renal replacement therapy
5. To assess the overall duration of vasoactive medication use
6. To assess toxicity and tolerability

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU within 12 hours of presentation to the emergency department for septic shock requiring 15-25 mcg/min of norepinephrine. Septic shock will be defined as having a known or presumed infection with two or more criteria of systemic inflammatory response syndrome, a mean arterial pressure <65 mm Hg despite fluid resuscitation requiring vasopressor support, and a serum lactate >2 mmol/L. Criteria of systemic inflammatory response syndrome include a temperature >100.4°F or <96.8°F; heart rate >90/min; respiratory rate >20/min and a white blood cell count >12,000/mm3 or <4,000/mm3.

Exclusion Criteria:

* Age <18 years
* Pregnancy or lactation
* Known allergic reactions to angiotensin-II or hydrocortisone sodium succinate
* Requiring >25 mcg/min of norepinephrine or on any vasopressor other than norepinephrine at study enrollment
* Clinically significant bleeding precluding the use of chemical prophylaxis for venous thromboembolism
* Treatment with another investigational drug or other intervention during study timeframe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of hemodynamic response, defined as a decrease in norepinephrine-equivalent dose with a MAP ≥65 mm Hg at 1 hour after initiation of angiotensin-II | 1 hour
  Defined as a decrease in norepinephrine-equivalent dose with a MAP ≥65 mm Hg at 1 hour after initiation of angiotensin-II.

SECONDARY OUTCOMES:
The incidence of hemodynamic response at 3 hours after initiation of angiotensin-II | 3 hours
  Defined as a decrease in norepinephrine-equivalent dose with a MAP ≥65 mm Hg at 3 hours after initiation of angiotensin-II.
The incidence of hemodynamic response at 6 hours after initiation of angiotensin-II | 6 hours
  Defined as a decrease in norepinephrine-equivalent dose with a MAP ≥65 mm Hg at 6 hours after initiation of angiotensin-II.
28-day mortality | 28 days
  Defined as all cause mortality up to 28 days from study enrollment.
ICU length of stay | 1 year
  Defined as the time spent within the ICU until discharge to a step down unit.
Need for renal replacement therapy | 1 year
  Defined as patients started on either continuous renal replacement therapy (CRRT) or intermittent hemodialysis (IHD) during the study period.
Vasoactive medication duration overall | 1 year
  Defined as the duration (hours) of vasoactive medication use during the study period.
Incidence of adverse reactions | 1 year
  Define as an unexpected or unintended effect suspected to be caused by a medicine.

CONTACTS AND LOCATIONS:
Overall Officials: Tyson Dietrich, PharmD, Principal Investigator — Kingman Regional Medical Center
Locations (1):
- Kingman Regional Medical Center, Kingman, Arizona, United States

IPD SHARING:
Plan to Share IPD: No